CLINICAL TRIAL: NCT07250126
Title: 3D Biomimetic Spine Unit Model Through the Integration of Bioprinting and Transcriptomics (CDP-SUBT)
Acronym: CDP-SUBT
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: CDP-SUBT; GR20250006 (Other: Fondazione CDP)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Degenrative Disc Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The general objective of this project is to define the transcriptional profile of primary human cells derived from the nucleus pulposus (NP), annulus fibrosus (AF), and cartilaginous endplate (CEP), and to use this information as a reference to assess the biological relevance of a biomimetic spinal unit model obtained through bioprinting. By developing an in vitro model of human origin that incorporates key components of the spinal unit and applying transcriptional analyses to both native cells and their counterparts recovered from the 3D construct, the study will evaluate how accurately the bioprinted model reproduces the identity and heterogeneity of the native discal environment.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the Informed Consent for the study
* Age 30-70 years (included)
* Pfirrmann grade III-V
* Need to undergo spinal surgery

Exclusion Criteria:

* Presence of HIV, HBC, HCV or TPHA infection

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient affected by Degenerative Disc disease undergoing spinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Discovery of Tissue-Specific Molecular Markers in Intervertebral Disc Cellular Populations | From enrollment to data analysis (24 months)
  To identify genes that are specifically upregulated in one of the three intervertebral disc cellular populations-nucleus pulposus (NP), annulus fibrosus (AF), and cartilaginous endplate (CEP)-through comparative gene expression analysis of paired samples obtained from the same donors. This aim seeks to determine tissue-specific molecular markers that will be subsequently applied to the characterization of bioprinted intervertebral disc models.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, MI, Italy